CLINICAL TRIAL: NCT06642935
Title: A Feasibility, Interventional, Prospective Study to Enhance Features and Optimise the Clinical Pathway for the TICI Research System in Adult Cochlear Implant Recipients
Brief Title: A Study to Explore Improved Features and a Simplified Treatment Approach for a Totally Implantable Cochlear Implant (TICI) Research System in Adults With Severe Hearing Loss
Acronym: ENHANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI5848; AI5848 (Other: Cochlear)
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hearing Loss, Bilateral or Unilateral; Hearing Loss, Sensorineural; Hearing Loss, Cochlear
Keywords: cochlear implant; sensorineural hearing loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device :TICI G2 Clinical Investigation System (Experimental): Totally implantable cochlear Implant
  Interventions: Device: Totally implantable cochlear Implant

INTERVENTIONS:
Device: Totally implantable cochlear Implant — Totally implantable cochlear Implant

SUMMARY:
This clinical study will test a new investigational totally implanted cochlear implant system (TICI G2). The cochlear implant has an implantable microphone under the skin to detect speech and sound from the environment allowing hearing without the need of any external parts. This study will explore new ways to process the sound from the implanted microphone. The study will be conducted in adults with sensorineural hearing loss, a type of hearing loss caused by damage to the inner ear or auditory nerve. The study participants will undergo a series of tests that include testing their implant and their hearing. They will also complete questionnaires to see how they rate their hearing and overall general health.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, at time of consent
* Candidate for cochlear implantation as assessed by the implanting clinic
* Fluent in English, as determined by the investigator
* Willing to participate in and comply with all requirements of the protocol
* Willing and able to provide written informed consent

Exclusion Criteria:

* Severe, or poorer, bilateral sensorineural hearing loss prior to five years of age, as reported by the subject
* Duration of severe to profound hearing loss greater than 20 years in the ear to be implanted as reported by the subject or by audiometric history, if available
* Ossification, otosclerosis, malformation or any other cochlear anomaly, such as common cavity, that might prevent complete insertion of the electrode array
* Deafness due to lesions of the acoustic nerve affecting the ear to be implanted
* Medical or psychological conditions that would contraindicate undergoing anaesthesia, surgery or participation in the clinical investigation, as determined by the investigator
* Additional disabilities that may affect the subject's participation or safety during the clinical investigation, as determined by the investigator
* Unrealistic expectations on the part of the subject regarding the possible benefits, risks and limitations that are inherent to the surgical procedure and prosthetic device, as determined by the investigator
* Desire to use an integrated acoustic component post-implantation
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling
* Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless Cochlear sponsored and determined by investigator or Sponsor to not impact this investigation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Mean change in the cochlear implant internal microphone frequency gain response over time | 1 day, 7 days, 14 days, 21 days, 8 weeks (60 days), 12 weeks (90 days), 52 weeks (12 months) and 77 weeks (18 months) post-implantation surgery
  The mean gain (dB) averaged across the frequency range (0.125 to 8kHz) of the internal cochlear implant microphone measured at 1 day, 7 days, 14 days, 21 days, 8 weeks (60 days), 12 weeks (90 days), 52 weeks (12 months) and 77 weeks (18 months) post-implantation surgery

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Moran, Study Director — Cochlear Ltd
Locations (1):
- Royal Victoria Eye and Ear Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No